CLINICAL TRIAL: NCT00617097
Title: Paracervical Block With Ketorolac and Lidocaine in First Trimester Surgical Abortions
Brief Title: Paracervical Block in First Trimester Surgical Abortions
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NA_00013075; SFP1-1 (Other Grant/Funding Number: Society of Family Planning)
Record Dates: First submitted 2007-12-28; First posted 2008-02-15 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-08

CONDITIONS: Pain; Surgical Abortion
Keywords: Pain associated with first trimester surgical abortion
MeSH Terms: conditions — Pain | interventions — Lidocaine; Ketorolac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- paracervical block with lidocaine (Active Comparator): Subjects who receive pain control using paracervical block with lidocaine during first trimester surgical abortion
  Interventions: Drug: lidocaine
- paracervical block with ketorolac and lidocaine (Experimental): Subjects who receive pain control using paracervical block with ketorolac and lidocaine during first trimester surgical abortion
  Interventions: Drug: ketorolac and lidocaine

INTERVENTIONS:
Drug: lidocaine — paracervical block with lidocaine
  Arms: paracervical block with lidocaine
Drug: ketorolac and lidocaine — paracervical block with ketorolac and lidocaine
  Arms: paracervical block with ketorolac and lidocaine

SUMMARY:
The investigators primary objective is to study the analgesic effects of combined ketorolac and lidocaine in a paracervical block compared to preoperative ibuprofen followed by intra-operative paracervical block with lidocaine alone on women undergoing first trimester surgical abortions. The investigators hypothesize that women who receive a paracervical block of combined ketorolac and lidocaine will experience less pain during the procedure based on a visual analog scale (VAS) compared to those who receive preoperative ibuprofen and a paracervical block with lidocaine alone.

This randomized, multi-site, placebo-controlled clinical trial will investigate the difference in perceived pain from first trimester surgical abortions using a paracervical block of combined ketorolac and lidocaine compared to preoperative ibuprofen and paracervical block with lidocaine alone. A total of fifty women who are seeking elective surgical abortions of intrauterine pregnancies less than 11 0/7 weeks' gestation will be recruited from Johns Hopkins Bayview Medical Center, Planned Parenthood of Maryland in Baltimore, Maryland and Planned Parenthood Columbia-Willamette in Portland, Oregon. Pain before, during, and after surgical abortion will be measured using a 100-mm VAS.

The primary outcome of interest is the mean difference in pain level from preoperative baseline to time after cervical dilation comparing the treatment groups. If the investigators see greater pain reduction associated with the paracervical block of lidocaine and ketorolac, adoption of this regimen may improve pain management during first trimester surgical abortions. If combined ketorolac and lidocaine when administered as a paracervical block is proven to be efficacious, the need for additional analgesia in first trimester surgical abortions can be minimized.

ELIGIBILITY:
Inclusion Criteria:

* age greater than or equal to 18 years
* English-speaking
* ability and willingness to sign the informed consent
* ability and willingness to comply with the terms of the study
* voluntary request for pregnancy termination
* ultrasound-confirmed singleton intrauterine pregnancy with an estimated gestational age not exceeding 76 days (10 6/7 weeks) from the first day of the preceding menstrual cycle

Exclusion Criteria:

* women who require or request sedation
* untreated acute cervicitis or pelvic inflammatory disease
* contraindications to lidocaine such as allergy to lidocaine, cardiac arrhythmia or heart block, and porphyria
* allergic reaction or sensitivity to lorazepam or NSAIDs
* chronic NSAID use
* history of gastritis or gastric ulcer
* acute renal failure or chronic renal disease
* chronic liver disease
* history of bleeding diathesis
* chronic narcotic use
* current or past history of illegal drug use (excluding marijuana)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2008-01; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johns Hopkins University, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Planned Parenthood Columbia-Willamette, Portland, Oregon, United States

REFERENCES:
- [Derived] Cansino C, Edelman A, Burke A, Jamshidi R. Paracervical block with combined ketorolac and lidocaine in first-trimester surgical abortion: a randomized controlled trial. Obstet Gynecol. 2009 Dec;114(6):1220-1226. doi: 10.1097/AOG.0b013e3181c1a55b. PMID 19935022

RESULTS

PARTICIPANT FLOW:
Groups:
- Paracervical Block With Lidocaine: Subjects who received paracervical block with 18 mL of 1% lidocaine and 2 mL of saline for pain control during first trimester surgical abortion
- Paracervical Block With Ketorolac and Lidocaine: Subjects who received pain control of paracervical block with combined 30mg of ketorolac and 18mL of 1% lidocaine during first trimester surgical abortion
Period: Overall Study
Arm/Group | Paracervical Block With Lidocaine | Paracervical Block With Ketorolac and Lidocaine
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Paracervical Block With Lidocaine: Subjects who received pain control with paracervical block with 18mL of 1% lidocaine and 2mL of saline during first trimester surgical abortion
- Paracervical Block With Ketorolac and Lidocaine: Subjects who received pain control with paracervical block with 30mg (2mL) of ketorolac and 18mL of 1% lidocaine during first trimester surgical abortion
- Total: Total of all reporting groups
Arm/Group | Paracervical Block With Lidocaine | Paracervical Block With Ketorolac and Lidocaine | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (6.2) | 25.6 (5.4) | 26.3 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 23 | 24 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 7 | 15
  White | 12 | 13 | 25
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50
gestational age [Mean (Standard Deviation); unit: days] | 54 (10.1) | 57.3 (11) | 55.7 (10.6)
gravidity [Number; unit: participants]
  1 | 6 | 9 | 15
  2 | 6 | 3 | 9
  3 | 5 | 2 | 7
  4 or greater | 8 | 10 | 18
  Missing data | 0 | 1 | 1
prior vaginal deliveries [Number; unit: participants]
  0 | 17 | 18 | 35
  1 or more | 8 | 7 | 15
prior abortions [Number; unit: participants]
  0 | 15 | 15 | 30
  1 or more | 10 | 9 | 19
  Missing data | 0 | 1 | 1
level of provider performing procedure [Number; unit: participants]
  resident/fellow | 9 | 7 | 16
  attending | 16 | 18 | 34
institution [Number; unit: participants]
  Johns Hopkins University | 14 | 14 | 28
  Oregon Health and Science University | 11 | 11 | 22
level of menstrual symptoms [Number; unit: participants]
  easy | 8 | 7 | 15
  mild cramping, no medications | 9 | 4 | 13
  over-the-counter medication use | 8 | 14 | 22

OUTCOME MEASURES:

1. Primary Outcome: Level of Pain During Specific Time Intervals Throughout D&C Procedure.
Description: 100-mm Visual Analogue Scale (VAS) during specific time intervals of D&C procedure: minimum: 0 mm (less pain); maximum: 100 mm (more pain)
  Time intervals include: basline expected level of pain during procedure, after speculum insertion, at paracervical block injection, after dilation, end of procedure, and 30 minutes after procedure.
Time Frame: Baseline, Speculum Insertion, at Paracervical block injection, After dilation, End of procedure, 30 minutes after procedure
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Paracervical Block With Lidocaine: Subjects who received pain control using paracervical block with 18mL of 1% lidocaine and 2 mL of saline during first trimester surgical abortion
- Paracervical Block With Ketorolac and Lidocaine: Subjects who received pain control using paracervical block with 30mg (2mL) of ketorolac and 18mL of 1% lidocaine during first trimester surgical abortion
Arm/Group | Paracervical Block With Lidocaine | Paracervical Block With Ketorolac and Lidocaine
Number analyzed (Participants) | 25 | 25
mm
  expected level of pain during procedure | 52.2 (20.8) | 51.7 (25.4)
  after speculum insertion | 33.6 (23.2) | 32.7 (26.6)
  during paracervical block administration | 50.8 (23.6) | 46.0 (24.3)
  after cervical dilation | 74.8 (19.0) | 59.8 (25.1)
  immediately after procedure | 61.5 (24.6) | 64.3 (27.4)
  30 min after procedure | 21.8 (22.4) | 17.6 (21.4)
Statistical Analysis 1: Comparison: Paracervical Block With Lidocaine vs Paracervical Block With Ketorolac and Lidocaine; expected level of pain during procedure greater number is worse (i.e., more pain) 100-mm Visual Analogue Scale (VAS): minimum: 0 mm (less pain); maximum: 100 mm (more pain); Test type: Superiority or Other; p = 0.94, Regression, Linear; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-13.7 to 12.6]
Statistical Analysis 2: Comparison: Paracervical Block With Lidocaine vs Paracervical Block With Ketorolac and Lidocaine; after speculum insertion greater number is worse (i.e., more pain) 100-mm Visual Analogue Scale (VAS): minimum: 0 mm (less pain); maximum: 100 mm (more pain); Test type: Superiority or Other; p = 0.9, Regression, Linear; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-15.1 to 13.2]
Statistical Analysis 3: Comparison: Paracervical Block With Lidocaine vs Paracervical Block With Ketorolac and Lidocaine; during paracervical block administration greater number is worse (i.e., more pain) 100-mm Visual Analogue Scale (VAS): minimum: 0 mm (less pain); maximum: 100 mm (more pain); Test type: Superiority or Other; p = 0.49, Regression, Linear; Mean Difference (Final Values) = -4.8, 95% CI 2-sided [-18.6 to 9]
Statistical Analysis 4: Comparison: Paracervical Block With Lidocaine vs Paracervical Block With Ketorolac and Lidocaine; after cervical dilation greater number is worse (i.e., more pain) 100-mm Visual Analogue Scale (VAS): minimum: 0 mm (less pain); maximum: 100 mm (more pain); Test type: Superiority or Other; p = 0.03, Regression, Linear; Mean Difference (Final Values) = -15, 95% CI 2-sided [-28.3 to -1.7]
Statistical Analysis 5: Comparison: Paracervical Block With Lidocaine vs Paracervical Block With Ketorolac and Lidocaine; immediately after procedure greater number is worse (i.e., more pain) 100-mm Visual Analogue Scale (VAS): minimum: 0 mm (less pain); maximum: 100 mm (more pain); Test type: Superiority or Other; p = 0.7, Regression, Linear; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [-12.2 to 18]
Statistical Analysis 6: Comparison: Paracervical Block With Lidocaine vs Paracervical Block With Ketorolac and Lidocaine; 30 min after procedure greater number is worse (i.e., more pain) 100-mm Visual Analogue Scale (VAS): minimum: 0 mm (less pain); maximum: 100 mm (more pain); Test type: Superiority or Other; p = .52, Regression, Linear; Mean Difference (Final Values) = -4.1, 95% CI 2-sided [-17 to 8.8]

2. Secondary Outcome: Visual Analogue Scale Regarding Satisfaction Level
Description: 100-mm Visual Analogue Scale -- minimum: 0 mm (lower satisfaction), maximum: 100 mm (greater satisfaction)
Time Frame: end of study (prior to clinic discharge)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Paracervical Block With Lidocaine | Paracervical Block With Ketorolac and Lidocaine
Number analyzed (Participants) | 25 | 25
mm | 62.9 (24.6) | 63.6 (28.1)
Statistical Analysis 1: Comparison: Paracervical Block With Lidocaine vs Paracervical Block With Ketorolac and Lidocaine; greater number is better (i.e., more satisfaction) 100-mm Visual Analogue Scale (VAS): minimum: 0 mm (less satisfaction); maximum: 100 mm (greater satisfaction) Measured at end of study (i.e., upon clinic discharge); Test type: Superiority or Other; p = 0.93, Regression, Linear

3. Secondary Outcome: Reported Symptoms
Description: fever, chills, vomiting, heavy bleeding/clots (collected without regard to the specific event)
Time Frame: end of study (upon discharge from facility after procedure)
Measure: Number; unit: participants
Arm/Group | Paracervical Block With Lidocaine | Paracervical Block With Ketorolac and Lidocaine
Number analyzed (Participants) | 25 | 25
participants | 3 | 0
Statistical Analysis 1: Comparison: Paracervical Block With Lidocaine vs Paracervical Block With Ketorolac and Lidocaine; greater number is worse (i.e., more symptoms); Test type: Superiority or Other; p = 0.07, Chi-squared

4. Secondary Outcome: Complications
Time Frame: end of study
Measure: Number; unit: participants
Arm/Group | Paracervical Block With Lidocaine | Paracervical Block With Ketorolac and Lidocaine
Number analyzed (Participants) | 25 | 25
participants
  minor | 1 | 1
  serious | 0 | 2
Statistical Analysis 1: Comparison: Paracervical Block With Lidocaine vs Paracervical Block With Ketorolac and Lidocaine; minor complications greater number is worse (i.e., more complications); Test type: Superiority or Other; p = 1, Chi-squared
Statistical Analysis 2: Comparison: Paracervical Block With Lidocaine vs Paracervical Block With Ketorolac and Lidocaine; serious complications; Test type: Superiority or Other; p = 0.15, Chi-squared

ADVERSE EVENTS:
Time Frame: Data collected during study participation (receipt of written informed consent until 2-4 week follow-up by phone or clinic visit)
Arm/Group | Paracervical Block With Lidocaine | Paracervical Block With Ketorolac and Lidocaine
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/25
Other Adverse Events (participants affected / at risk) | 3/25 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paracervical Block With Lidocaine (N=25) | Paracervical Block With Ketorolac and Lidocaine (N=25)
immediate postoperative hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) — Subject experienced hemorrhage (400mL) most likely due to subject's known leiomyoma. Subject was treated conservatively as an outpatient and did not require blood transfusion.
repeat procedure (Reproductive system and breast disorders) | 0 (0) | 1 (1) — Subject underwent uncomplicated repeat vacuum aspiration procedure on postoperative day 3.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paracervical Block With Lidocaine (N=25) | Paracervical Block With Ketorolac and Lidocaine (N=25)
reported symptoms (Reproductive system and breast disorders) | 3 (3) | 0 (0) — Secondary outcomes assessed included fever, chills, vomiting, heavy bleeding/clots.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No